CLINICAL TRIAL: NCT06435039
Title: A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of APL-1501 ER Capsules Compared to APL-1202 IR Tablets in Healthy Volunteers
Brief Title: A Study of APL-1501 Extended Release Capsules Compared to APL-1202 Immediate Release Tablets in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated by sponsor due a business decision and development strategy.
Sponsor: Syneos Health (Other)
Collaborators: Asieris Pharmaceuticals (AUS) Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHGT-APL1501-NHS-103
Record Dates: First submitted 2024-05-22; First posted 2024-05-30 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1, Sequence 1, R1T1: APL-1202 IR 375 mg + APL-1501 ER 764 mg (Experimental): Participants will receive APL-1202 375 milligram (mg) IR tablets, orally, once on Day 1 of Period 1 (Treatment R1), followed by T1 APL-1501 764 mg ER capsules, orally, once, on Day 4 of Period 2 (Treatment T1). A washout period of more than or equal to (>=) 72 hours will be maintained in between Period 1 and 2.
  Interventions: Drug: APL-1202; Drug: APL-1501
- Cohort 1, Sequence 2, T1R1: APL-1501 ER 764 mg + APL-1202 IR 375 mg (Experimental): Participants will receive APL-1501 764 mg ER capsules, orally, once on Day 1 of Period 1 (Treatment T1), followed by APL-1202 375 mg IR tablets, orally, once, on Day 4 of Period 2 (Treatment R1). A washout period of >=72 hours will be maintained in between Period 1 and 2.
  Interventions: Drug: APL-1202; Drug: APL-1501
- Cohort 2, Sequence 1, R1T2: APL-1202 IR 375 mg + APL-1501 ER 1146 mg (Experimental): Participants will receive APL-1202 375 mg IR tablets, orally, once on Day 1 of Period 1 (Treatment R1), followed by APL-1501 1146 mg ER capsules, orally, once, on Day 4 of Period 2 (Treatment T2). A washout period of >=72 hours will be maintained in between Period 1 and 2.
  Interventions: Drug: APL-1202; Drug: APL-1501
- Cohort 2, Sequence 2, T2R1: APL-1501 ER 1146 mg + APL-1202 IR 375 mg (Experimental): Participants will receive APL-1501 1146 mg ER capsules, orally, once on Day 1 of Period 1 (Treatment T2), followed by APL-1202 375 mg IR tablets, orally, once, on Day 4 of Period 2 (Treatment R1). A washout period of >=72 hours will be maintained in between Period 1 and 2.
  Interventions: Drug: APL-1202; Drug: APL-1501
- Cohort 3: APL-1501 ER 1528 mg (Experimental): Participants will receive APL-1501 1528 mg ER capsules, orally, once on Day 1.
  Interventions: Drug: APL-1501

INTERVENTIONS:
Drug: APL-1202 — APL-1202 IR tablets.
  Arms: Cohort 1, Sequence 1, R1T1: APL-1202 IR 375 mg + APL-1501 ER 764 mg; Cohort 1, Sequence 2, T1R1: APL-1501 ER 764 mg + APL-1202 IR 375 mg; Cohort 2, Sequence 1, R1T2: APL-1202 IR 375 mg + APL-1501 ER 1146 mg; Cohort 2, Sequence 2, T2R1: APL-1501 ER 1146 mg + APL-1202 IR 375 mg
Drug: APL-1501 — APL-1501 ER capsules.

SUMMARY:
The primary objective of the study is to assess safety and tolerability following administration of single doses of APL-1202 (immediate release) IR tablets and APL-1501 extended release (ER) capsules in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in the study:

1. Male, >=18 and less than or equal to (<=) 65 years of age, with body mass index (BMI) greater than (>) 18.5 and less than (<) 32.0 kilogram per square meter (kg/m^2) and body weight >=50.0 kilogram (kg).
2. Non-smoker (no use of tobacco or nicotine products, example, snuff, chewing tobacco, cigars, cigarettes, pipes, e-cigarettes [vaping] etc. within 3 months prior to screening).
3. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to study drug administration.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
4. Sexually active non-sterile males must be willing to use an acceptable contraceptive method throughout the study.
5. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

Participants to whom any of the following applies will be excluded from the study:

1. Any clinically significant abnormal finding at physical examination.
2. Clinically significant abnormal laboratory test results or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV) antibody, or Human immunodeficiency virus (HIV) antigen and antibody.
3. Positive urine drug screen, cotinine test, or alcohol breath test.
4. History of significant allergic reactions (example, anaphylactic reaction, hypersensitivity, angioedema) to any drug.
5. Clinically significant Electrocardiograms (ECG) abnormalities or vital signs abnormalities (systolic blood pressure [BP] lower than 90 or over 140 millimeters of mercury [mmHg], diastolic BP lower than 50 or over 90 mmHg, heart rate [HR] less than 40 or over 100 beats per minute [bpm], or RR less than 10 or over 25 bpm) at screening.
6. History of drug abuse within 1 year prior to screening or recreational use of marijuana within 1 month or other illegal drugs such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives within 3 months prior to screening.
7. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units of alcohol per week (1 unit = 375 milliliter [mL] of beer 3.5 percent (%), or 100 mL of wine 13.5%, or 30 mL of distilled alcohol 40%).
8. Use of medications within the timeframes specified in section.
9. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
10. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
11. Optic nerve disease, cataracts, or a history of related conditions.
12. Any reason which, in the opinion of the Investigator, would prevent the participant from participating in the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | From Baseline up to Day 9
Number of Participants With Abnormal Vital Sign Measurements | From Baseline up to Day 9
Number of Participants With Abnormal 12-Lead Electrocardiogram (ECGs) Recordings | From Baseline up to Day 9
Number of Participants With Abnormal Physical Examinations | From Baseline up to Day 9
Number of Participants With Abnormal Clinical Laboratory Values | From Baseline up to Day 9

SECONDARY OUTCOMES:
AUC0-t: Area Under the Concentration-time Curve From Time Zero Until the Last Observed Concentration of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
AUC0-inf: Area Under the Concentration-time Curve From Time Zero to Infinity of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Cmax: Maximal Observed Concentration of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Tlast: Time When the Last Concentration is Observed of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Tmax: Time When the Cmax is Observed of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Residual Area of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
  Residual area is defined as percentage of AUC0-inf due to extrapolation from the time of the last observed concentration to infinity and is calculated as, [1-(AUC0-t/AUC0-inf)]*100.
T½ el: Terminal Elimination Half-life of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Kel: Terminal Elimination Rate Constant of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Cl/F: Apparent Clearance of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Vz/F: Apparent Volume of Distribution of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
DNAUC0-inf: Dose Normalized AUC0-inf of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
DNCmax: Dose Normalized Cmax of APL-1202, and ASN-1651 (Metabolite) Following APL-1501 ER Capsules | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Geometric Mean Ratio of Cmax of APL-1501 ER Capsules in Reference to APL-1202 IR Tablets | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Geometric Mean Ratio of AUC0-t of APL-1501 ER Capsules in Reference to APL-1202 IR Tablets | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Geometric Mean Ratio of AUC0-inf of APL-1501 ER Capsules in Reference to APL-1202 IR Tablets | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
Frel: Relative Bioavailability of APL-1501 ER Capsules and APL-1202 IR Tablets | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
  The relative bioavailability of APL-1501 versus APL-1202 will be assessed through linear mixed modelling.
Dose Proportionality of Cmax | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
  Dose proportionality will be assessed by visual inspection of dose normalised Cmax values versus dose.
Dose Proportionality of AUC0-t | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
  Dose proportionality will be assessed by visual inspection of dose normalised AUC0-t values versus dose.
Dose Proportionality of AUC0-inf | Cohorts 1 and 2 - Days 1 and 4: Pre-dose and up to 24 hours post-dose; Cohort 3 - Day 1: Pre-dose and up to 24 hours post-dose
  Dose proportionality will be assessed by visual inspection of dose normalised AUC0-inf values versus dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Christopher Argent, Principal Investigator — Asieris Pharmaceuticals (AUS) Pty Ltd.
Locations (1):
- Scientia Clinical Research Ltd, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No